CLINICAL TRIAL: NCT02570633
Title: Double-blind Placebo-controlled Clinical Trial of Ginger (Zingiber Officinale) in Prophylactic Migraine Treatment
Brief Title: Ginger Capsules for the Prophylactic Treatment of Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio L Teixeira Jr, PhD, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CAAE 28236814.3.0000.5149
Record Dates: First submitted 2015-10-02; First posted 2015-10-07 (Estimated); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Migraine
Keywords: Migraine; Ginger; Prophylactic treatment
MeSH Terms: conditions — Migraine Disorders | interventions — Cellulose

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extract of ginger (Experimental): Migraine patients (both genders) will receive capsules of 200 mg of ginger extract (5% gingerols) to be taken three times a day for 12 weeks.
  Interventions: Other: Extract of ginger
- Cellulose (Placebo Comparator): Migraine patients (both genders) will receive capsules of 200 mg of placebo (cellulose) to be taken three times a day for 12 weeks.
  Interventions: Other: Cellulose

INTERVENTIONS:
Other: Extract of ginger — Migraine patients (both genders) will receive capsules of 200 mg of ginger extract (5% gingerols) to be taken three times a day for 12 weeks.
  Arms: Extract of ginger
Other: Cellulose — Migraine patients (both genders) will receive capsules of 200 mg of placebo (cellulose) to be taken three times a day for 12 weeks.
  Arms: Cellulose

SUMMARY:
The main objective of the study is to evaluate ginger efficacy as an prophylactic treatment of migraine.

DETAILED DESCRIPTION:
Patients with the diagnosis of migraine according to the IHS criteria will receive capsules of 200 mg of ginger extract (5% active ingredient) or placebo (cellulose) to be taken three times a day for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60 years old;
* Migraine diagnosis;
* Agree to sign the informed consent.

Exclusion Criteria:

* Patients with headaches not characterized as migraine;
* Pregnant or lactating women;
* Fertile and sexually active women who do not use contraception;
* Abuse of painkillers, alcohol or other drugs;
* People with hypersensitivity to ginger compounds;
* People with severe neurological diseases (e.g. epilepsy)
* People in use of anticoagulant drugs.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in the frequency of migraine attacks. | 12 weeks
  Frequency of migraine attacks will be assessed by headache diary.

SECONDARY OUTCOMES:
Change in migraine impact in the last month. | 4 weeks
  Migraine impact will be assessed by HIT-6.
Change in migraine impact in the last three months. | 12 weeks
  Migraine impact will be assessed by MIDAS.
Changes in the serum levels of biomarkers. | 12 weeks
  Biomarkers: inflammatory mediators and neurotrophic factors
Changes in Resting Energy Expenditure | 4, 8 and 12 weeks
  Resting Energy Expenditure will be assessed by calorimeter

CONTACTS AND LOCATIONS:
Overall Officials: Adaliene VM Ferreira, PhD, Study Director — Federal University of Minas Gerais; Laís B Martins, Ma, Study Chair — Federal University of Minas Gerais; Antônio L Teixeira, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Ambulatório Bias Fortes, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Martins LB, Rodrigues AMDS, Monteze NM, Tibaes JRB, Amaral MHA, Gomez RS, Teixeira AL, Ferreira AVM. Double-blind placebo-controlled randomized clinical trial of ginger (Zingiber officinale Rosc.) in the prophylactic treatment of migraine. Cephalalgia. 2020 Jan;40(1):88-95. doi: 10.1177/0333102419869319. Epub 2019 Aug 9. PMID 31398997